CLINICAL TRIAL: NCT01702792
Title: Vaccination of Patients With Newly Diagnosed Glioblastoma Using Autologous Tumor Lysate and Montanide Emulsion for Derivation of Tumor Specific Hybridomas
Brief Title: Derivation of Tumor Specific Hybridomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator is leaving Dartmouth
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: University of Vermont (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W12209
Record Dates: First submitted 2012-10-03; First posted 2012-10-08 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Glioblastoma
Keywords: Immunotherapy, cancer vaccine, glioblastoma, hybridoma
MeSH Terms: conditions — Glioblastoma | interventions — Cancer Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tumor Vaccine (Experimental): 1 x 107 TCE tumor lysate in 0.5 ml Lactated Ringers Solution (approximately 1 mg of tumor lysate protein) and equivalent volume of adjuvant will be injected 2 weeks and 3 weeks (2 vaccinations) after surgery in the intradermal skin of the upper thigh. There will be 2 vaccine administrations and patients will be followed for 2 months after inguinal node removal for any possible vaccine/study-related toxicity.
  Interventions: Biological: Tumor Vaccine

INTERVENTIONS:
Biological: Tumor Vaccine — Tumor cells obtained at the time of surgery are irradiated with 10,000 Gy and freeze fractured. Lysate at 1x107 tumor cell equivalent (TCE) will be used for vaccination with adjuvant, Montanide ISA 51 VG.
  Other Names: Autologous Tumor Lysate and Montanide Emulsion

SUMMARY:
This is a non-randomized, open-label study in patients with newly diagnosed glioblastoma to determine the ability to generate human hybridomas from lymph nodes draining an autologous tumor vaccine injection and demonstrate that the hybridomas secrete glioblastoma-specific antibodies.

DETAILED DESCRIPTION:
The intradermal vaccine will be injected 20cm in the anterior thigh. Vaccination will be done twice and separated by one week. The first vaccination will be performed approximately 2 weeks after surgery.

Approximately one week after the second vaccination one or two vaccine-draining lymph node(s) will be removed. The lymph node(s) will be identified using SN technology. One or two lymph node(s) will be removed.

Lymph nodes will be processed for recovery of B cells and formation of hybridomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed new diagnosis of glioblastoma and who have a yield of at least 8x10(7) tumor cells obtained at the time of surgery
* Age > 18 years
* KPS Score of greater than or equal to 70
* Adequate bone marrow as evidenced by:

Absolute lymphocyte count > 1,000/uL Platelet count > 50,000/uL

* Adequate renal function as evidenced by serum creatinine < 2.0
* Patients must be able to read, understand and provide informed consent to participate in the trial.
* Patients of childbearing potential must agree to use an effective form of contraception during the study and for 90 days following vaccination (an effective form of contraception is an oral contraceptive or a double barrier method)

Exclusion Criteria:

A patient may not be enrolled in the trial if any of the following criteria are met:

* Patients receiving dexamethasone > 8 mg/day during the week before vaccination.
* Patients who are pregnant or lactating
* Patients with active second malignancy.
* Any other medical conditions, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05-06 (Actual); Study Completion 2015-05-06 (Actual)

PRIMARY OUTCOMES:
number of hybridoma clones that produce anti-glioma antibodies | 6 months
  The primary technical endpoint demonstrating the feasibility of the pilot study will be based upon the total count of the number of generated hybridoma clones sourced from the dermal vaccine draining lymph nodes that are determined to be producing anti-glioma antibodies.

SECONDARY OUTCOMES:
Production of Antibodies | 6 months
  Secondary outcomes will include:
  Determining how many hybridoma clones produce glioblastoma-specific antibodies. The initial secondary endpoint will include the counting of the number of hybridoma clones sourced from the dermal vaccine draining lymph nodes that generate specific glioma antibodies.
Toxicity of Vaccine | 6 months
  • Determining toxicity of vaccine
Clone Production Rate | 6 months
  Determining whether B cells sourced from the vaccine nodes produce more anti-tumor antibody hybridomas than the non-vaccine node. The rate of producing these clones will be compared according to the source of the B cells. Thus, B cells recovered from vaccine related nodes will be compared to B cells recovered from the non-vaccine node.
Lymph Node Biopsy | 6 months
  Determine the safety and toxicity issues related to the Lymph Node Biopsy

OTHER OUTCOMES:
Tumor Binding Characteristics | 6 months
  Exploratory objectives will include:
  * Determining the rate of tumor binding antibodies from hybridomas derived from circulating B cells.
  * Determining the tumor-binding profile of antibodies present in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Fadul, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center